CLINICAL TRIAL: NCT05607407
Title: Targeting Transsulfuration Via Suppression of Thyroid Hormone Signaling in Progressive Glioblastoma: Phase 2 and Pharmacodynamic Trial of Methimazole in Patients With Progressive Glioblastoma
Brief Title: Methimazole in Patients With Progressive Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3322
Record Dates: First submitted 2022-10-26; First posted 2022-11-07 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Glioma
Keywords: Transsulfuration; Methimazole
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Methimazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Surgical Resection, Pharmacodynamic Assays, and Methimazole (Experimental): Participants with recurrent glioblastoma for whom surgical resection is indicated will have baseline peripheral blood pharmacodynamic assays (PBPD) followed by oral mehimazole at least 5 days pre-operatively or until lower circulating theyroid hormone levels are achieved. PBPD assays will then be repeated. After surgical resection, PBPD will be repeated a day later. When the participant is deemed able to begin methimazole (no sooner than 10 days post-op) PBPD assays will be repeated and the participant will begin methimazole for 4 weeks. At the end of the first 4 week cycle, an MRI will be performed. PBPD assays will be repeated after which secondary chemotherapy will be added at the treating physician's discretion. After 4 weeks, PBPD will be repeated and the participant will undergo another MRI at 8 weeks.
  Interventions: Drug: Methimazole; Procedure: Recurrent Glioblastoma Surgical Resection; Diagnostic Test: Pharmacodynamic Assays

INTERVENTIONS:
Drug: Methimazole — Starting dose: Methimazole 15 mg/d. Six participants will receive this dose. If they achieve a 10% increase in peripheral blood H2S concentrations, an additional 13 participants will receive this dose to accrue a total of 19 participants for which a preliminary estimate of PFS6 can be calculated. If the first 6 participants do not achieve a 10% increase in peripheral blood H2S concentrations, the dose will be increased to the second and final dose level of 25 mg/d at which 19 participants will be treated.
  Other Names: Northyx; Tapazole
Procedure: Recurrent Glioblastoma Surgical Resection — The purpose of resection is to remove as much tumor as possible to alleviate mass effect and to obtain brain tissue for experimental analysis.
Diagnostic Test: Pharmacodynamic Assays — Pharmacodynamic assays are intended to investigate drug and downstream drug-induced effects.

SUMMARY:
The purpose of this study is to test the effectiveness, safety, and tolerability of a drug called Methimazole. The investigational drug, Methimazole is not FDA approved for brain tumors, but it is used to treat thyroid illnesses. Different doses of Methimazole will be given to several study participants with glioblastoma. The first several study participants will receive the lowest dose. If the drug does not cause serious side effects, it will be given to other study participants at a higher dose. The doses will continue to increase for every group of study participants until the side effects occur that require the dose to be lowered. The procedures in this study are research blood draws, physical exams, collection of medical history, MRI scans, and study drug administration.

DETAILED DESCRIPTION:
Hydrogen sulfide (H2S), a by-product of cysteine metabolism, inhibits the growth of cultured glioblastoma cells and impairs progression of glioblastoma tumors developing in vivo in laboratory mice. Additionally, endogenous H2S production and signaling via protein sulfhydration are decreased in human glioblastoma brain tissues compared to non-cancerous brain tissue. Thus, boosting H2S levels is a promising and novel therapeutic strategy for treating glioblastoma. The use of exogenous H2S is difficult to translate to the clinic due to toxicity and volatility. Therefore, bolstering endogenous H2S synthesis and signaling represents a safe and promising method to mitigate disease progression. Based on previously published data, which detailed the use of the thyroid hormone inhibitor propylthiouracil (PTU) to enhance endogenous H2S production in mice, and a previous clinical trial at CCF utilizing PTU to increase the survival of glioblastoma patients, revisiting the use of thyroid hormone inhibitors to de-repress endogenous H2S production concurrent with standards of care poses a novel therapeutic avenue. In the nearly two decades since the aforementioned clinical trial, PTU has been largely replaced in clinical endocrinology by the safer and more efficient thyroid inhibitor methimazole. Given our recent success elucidating the importance of tumor suppressive H2S in the realm of GBM, it is hypothesized that reduced thyroid hormone production via oral methimazole intake will bolster the effectiveness of frontline therapy and extend survival by boosting H2S production and function within the tumor-bearing brain. The goal of this trial is to provide proof of the concept that suppression of thyroid hormone signaling via methimazole and subsequent augmentation of H2S synthesis and signaling is feasible in patients with glioblastoma. Achievement of this goal will motivate and guide further therapeutic development of this combinatorial therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed WHO grade 4 glioma (including tumors with molecularly defined grade 4 astrocytoma) for which a clinically indicated tumor resection is planned.
* Subjects must not have received methimazole for this disease.
* Age is greater than or equal to 18 years of age
* Performance status: Karnofsky Performance status ≥ 70%
* Subjects must have adequate organ function and laboratory parameters within 21 days of study entry as defined below: Hemoglobin ≥ 8 g/dl, Absolute neutrophil count ≥ 1,200/mcL, Platelet count ≥ 75,000/mcL, Total bilirubin < 1.5 x institutional upper limit of normal (ULN), AST (SGOT) ≤ 3 X institutional ULN, ALT (SGPT) ≤ 3 X institutional ULN, Calculated creatinine clearance > 50 mL/min, Prothrombin time/international normalized ratio (PT/INR) <1.4 for patients not on warfarin, Patients on full-dose anticoagulants (e.g., warfarin or LMW heparin) must meet both of the following criteria: No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices), In-range INR (between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
* Subjects must have normal thyroid function within 21 days of study entry as defined below: ≤ 3 X institutional ULN
* Women of childbearing potential must have a negative pregnancy test within 21 days of study entry. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 30 days after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Men of reproductive potential treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 30 days after the last dose of study drug.
* Patients must be able to swallow whole tablets.
* Patients must have the following minimum intervals from prior treatments: surgery - 4 weeks, nitrosoureas - 6 weeks, cytotoxic chemotherapy - standard intervals depending on the most recent regimen. i.e., for temozolomide 5 of 28, 23 days after most recent temozolomide; for temozolomide 21 of 28 days, 7 days after most recent dose; etoposide 14 of 21 days, 7 days after last dose. For drugs not listed, the research nurse, treating investigator, and principal investigator will determine the appropriate interval, Investigational therapy or non-cytotoxic therapy - 2 weeks, For bevacizumab - 4 weeks from anticipated date of protocol surgery
* Patients positive for human immunodeficiency virus (HIV) are allowed on study (note: HIV testing is not required), but HIV-positive patients must have: An undetectable viral load within 6 months of registration, A stable regimen of highly active anti-retroviral therapy (HAART), No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* For patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patient must be deemed by investigator to be a candidate for post-operative chemotherapy.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment toxicities not resolved to ≤ Grade 1 according to NCI CTCAE Version 5.0 except alopecia and neuropathy.
* Subjects receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to methimazole.
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Other prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are excluded. Otherwise, patients with prior or concurrent malignancy are eligible.
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or Grade ≥2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 5.0 [CTCAE v.5.0] diarrhea of any etiology at screening).
* Pregnant or breastfeeding.
* Known history of hyperthyroidism or hypothyroidism
* Unable or unwilling to swallow tablets.
* Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that would, in the Investigator's judgment, make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) Rate | Up to 6 months after treatment
  defined as alive and free from progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: David Peereboom, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States